CLINICAL TRIAL: NCT03854851
Title: NALDEBAIN for Postoperative Pain Management in Take Down of Anastomosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hung-Chang Chen, Director of Minimally Invasive Centre, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC2-110
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Postoperative Pain
Keywords: Naldebain; long-term analgesia; take down of anastomosis
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NALDEBAIN (Experimental): In group NALDEBAIN, subjects will receive single dose of Naldebain (150 mg/2 ml) by gluteus maximus injection between 12 and 24 hours prior to surgery.
  Interventions: Drug: Naldebain
- MORPHINE (Active Comparator): In group MORPHINE, subjects will receive morphine as needed after surgery.
  Interventions: Drug: Morpine

INTERVENTIONS:
Drug: Naldebain — In Naldebain group, patients will be injected with Naldebain (150 mg/2 ml, IM injection) between 12 and 24 hours prior to surgery.
  Arms: NALDEBAIN
Drug: Morpine — In Morphine group, patients will receive morphine as needed after surgery.
  Arms: MORPHINE

SUMMARY:
NALDEBAIN ER injection, invented by Taiwanese, launched in 2017, is a nalbuphine synthetic prodrug with oil-based solution to extend the release in human body by intramuscular injection. It was approved for the premedication use for moderate to severe pain relief, expected after surgery. There was limited experience with the combination of medication and different type of surgeries. Only the effect of operative analgesia on the hemorrhoidectomy patients have been well studied. Through reviewing the past medical cases, the pain intensity after receiving take down of anastomosis was about 4 to 7 points (moderate pain), lasing about 1 to 3 days. It was a suitable population with multi-day analgesic unmet need.

At present, the standard treatment after take down of anastomosis in the CMUH was morphine as needed. This treatment might not provide for well-controlled postoperative pain management. Patients might receive more painkillers when they needed than before pain occurred. Plus, it also cost more postoperative medical care. Therefore, this study intended to compare the standard treatment and NALDEBAIN for postoperative outcomes, safety and satisfaction.

The study will enroll patients scheduled to electively undergo take down of anastomosis. Eligible subjects were randomly divided into two groups, one receiving NALDEBAIN and the other receiving standard treatment. The study will evaluate pain intensity, dosage of supplement analgesics, incidence of adverse reactions, patient satisfaction, time of the first fart after surgery, and duration of postoperative hospital stay.

DETAILED DESCRIPTION:
This is an open-labeled, randomized clinical trial. After ICFs are signed, patients' medical history will be gained for checking if they are eligible for this study or not. And then, on Day -1, eligible ones will randomly be divide into two separate group: NALDEBAIN or MORPHINE. Group NALDEBAIN will receive Nadebain by gluteus maximus injection between 12 and 24 hours prior to surgery for postoperative pain relief. Group MORPHINE will receive morphine as needed after surgery. All necessary data will be gain form EMR or patient dairies.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women between 20 and 80 years of age
2. History of laparoscopic surgery
3. American Society of Anesthesiology Physical Class 1-3
4. Ability and willingness to provide informed consent

Exclusion Criteria:

1. History of hypersensitivity or allergy to opioid, NSAIDs, or Acetaminophen
2. Chronic preoperative opioid use
3. Severe comorbidity which is able to interfere pain assessment
4. Ostomy surgery of intestine within the past 8 weeks
5. Pregnant or breastfeeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Supplemental analgesics | From Day 0 to Day 7
  The consumption of total amount (mg) of supplemental analgesics administered after surgery.

SECONDARY OUTCOMES:
Pain assessment: VAS | 2 hours after surgery
  Using visual analog scale (VAS) with grades from 0 (no pain) to 10 (worst pain)
Pain assessment: VAS | 6 hours after surgery
  Using visual analog scale (VAS) with grades from 0 (no pain) to 10 (worst pain)
Pain assessment: VAS | 24 hours after surgery
  Using visual analog scale (VAS) with grades from 0 (no pain) to 10 (worst pain)
Pain assessment: VAS | From Day 2 to Day 7
  Using visual analog scale (VAS) with grades from 0 (no pain) to 10 (worst pain), once daily
Pain assessment: area under the curve of VAS | From post-OP to Day 7
  Pain assessment (time-specific pain intensity) calculated as the area under the curve of VAS pain intensity scores through 7 days after surgery
Patient satisfaction: frequency of each option | Day 7
  Calculating the frequency of each option: highly satisfied, satisfied, uncertain, dissatisfied and very dissatisfied
frequency of adverse event | From Day-1 to Day 7
  Recording the frequency of treatment-emergent adverse event (TEAE)

OTHER OUTCOMES:
Time of first farting | From post-OP to Day 7
  Observing when patients are able to pass gas after surgery
Date of discharge | From post-OP to Day 7
  Observing when the condition of patients is good enough to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chang Chen, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University & Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No